CLINICAL TRIAL: NCT06593535
Title: Short-term Astaxanthin Supplementation Enhances Cycling Performance and Attenuates Exhaustive Exercise-induced Muscle Damage and Oxidative Stress in Young Healthy Adults: A Randomized Controlled Trial
Brief Title: Evaluation of Astaxanthin Properties on Anti-fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); China Medical University, China (Other)
Responsible Party: Principal Investigator, Jung-Piao Tsao, Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CMUH111-REC3-081
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer
Keywords: Cycling performance; fatigue; ergogenic aids; lipid peroxidation
MeSH Terms: conditions — Fatigue | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Ten young healthy physically active male college students. Participants were crossed over for AST or placebo supplements, which was completed in four days. Between the crossover trials, participants had a one-week washout period to nullify the effects of the supplement
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): containing edible yellow No. 4, edible yellow No. 5, sucrose, silica, talc, oxidized starch, gelatin, magnesium stearate, and palm wax.
  Interventions: Other: Placebo (Placebo trial); Other: Astaxanthin (AST trial)
- Astaxanthin (AST) (Experimental): Each capsule containing 4 mg of AST
  Interventions: Other: Placebo (Placebo trial); Other: Astaxanthin (AST trial)

INTERVENTIONS:
Other: Placebo (Placebo trial) — The Placebo capsule supplement was taken for 4 days (7 capsules per day)
Other: Astaxanthin (AST trial) — The AST capsule supplement was taken for 4 days, with a daily dosage of 28 mg of AST (equivalent to 7 capsules per day, each containing 4 mg of AST).

SUMMARY:
Ten young, healthy, physically active male college students were crossed over for AST or placebo supplements randomized into placebo or AST trials and orally consumed placebo or AST (28 mg/d) supplements for four days. Short-term AST supplementation enhanced endurance performance and effectively reversed cycling challenge-induced muscle damage and lipid peroxidation.

DETAILED DESCRIPTION:
AST is composed of two β-ionone ring systems that are linked by a polyene chain and contain oxygenated keto and hydroxyl moieties, which are responsible for its powerful antioxidant activity. AST has been shown to have numerous health benefits in humans, including improved antioxidant and inflammatory status under different stress conditions. Therefore, this study will explore AST supplement to improve exercise-induced muscle damage and/or physiological anomalies in adults. Ten physically active male adults were randomized into placebo or AST trials and consumed placebo or AST (28 mg/d) supplements orally for 4 days. On day-4, participants performed an exhaustive cycling challenge at 75% V̇O2max, and the time to exhaustion (TTE) was recorded. Blood and gaseous samples were collected before, during, and immediately after cycling to determine changes in muscle damage, inflammation, oxidative stress, and substrate utilization.

ELIGIBILITY:
Inclusion Criteria:

* Recruit people who are healthy are 20-40 years male and have exercise habits in college students

Exclusion Criteria:

* Have smoking and drinking habits.
* Those who have implanted artificial joints in the past six months and have had recent surgery.
* People who feel unwell due to other reasons during the experiment.
* Take any drugs or Nutrition supplements in the past 3 months.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Time to Exhaustion Exercise | 21 days
  Investigators conducted a double-blind test, where volunteers' basal maximal oxygen consumption (VO2max) was measured both before the intervention. The pretest VO2max is a reference to adjust the exercise intensity for each individual. To assess exhaustive endurance, participants exercised at 75% of their VO2max, and the cycling time from the start to the point of exhaustion was recorded.
Clinical Biochemistry of muscle damage biomarkers and blood glucose | 21 days
  Blood samples were collected at five different time points (one hour before (B), at the beginning (0 min), during (20 min, 40 min), and immediately (E) after the exhaustive cycling exercise challenge. Changes in blood glucose levels were estimated using blood from the fingertips via an Accu-Chek® Guide blood glucose glucometer (Roche, Mannheim, Germany). Muscle damage biomarkers, including creatine kinase (CK), lactate dehydrogenase (LDH), and uric acid (UA), were measured in the serum. The CK (EC2.7.3.2), LDH (EC 1.1.1.27), and UA (C97792) concentrations were estimated using commercial analytical reagents (Beckman Coulter). An automated clinical chemistry analyzer was used to measure CK and LDH levels on a Beckman Coulter AU5800 (Beckman Coulter Inc., CA, USA).
Clinical Biochemistry of total antioxidant capacity and lipid peroxidation | 21 days
  Blood samples were collected at five different time points (one hour before (B), at the beginning (0 min), during (20 min, 40 min), and immediately (E) after the exhaustive cycling exercise challenge. The scavenging ability of antioxidants (6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid, Trolox) was determined using a curve, and the amount of Trolox equivalent to the test serum's inhibition rate was calculated. Next, the level of malondialdehyde (MDA), a standard biomarker of lipid peroxidation, was determined by an ELISA kit provided by the Caman Company (Cayman Chemical Company, Michigan, USA). As described in the protocol, the reaction mixture was boiled at 90-100°C for 60 min, and the absorbance at 550 nm was measured using an ELISA plate reader (Tecan GENios, A-5082, Austria). The values are expressed as micromoles of MDA per liter.
Clinical Biochemistry of the inflammatory response | 21 days
  Blood samples were collected at five different time points (one hour before (B), at the beginning (0 min), during (20 min, 40 min), and immediately (E) after the exhaustive cycling exercise challenge. According to the manufacturer's instructions, the pro-inflammatory cytokine TNF-α was analyzed with a commercial ELISA kit (BioLegend, San Diego, CA). An enzyme immunoassay read The absorbance at 450 nm within 15 minutes (Tecan GENios, A-5082, Austria). Concentrations of C-reactive protein (CRP) were measured using a human ELISA kit (E-80CRP, Immunology Consultants Laboratory, Inc., Newberg, OR, USA). The sample absorbance was read at 450 nm within 30 min.
Assessment of the profile of mood state (POMS) | 21 days
  POMS brief was chosen for this study to evaluate the mood of individuals. After the TTE, participants completed the form, and their responses were analyzed using simple statistics. The results were shown in six dimensions, one positive: (1) vigor; and five negatives: (2) tension, (3) depression, (4) anger, (5) fatigue and (6) confusion.
Assessment of the RER, fat oxidation rate and carbohydrate oxidation rate | 21 days
  Ggaseous samples were collected at five different time points (one hour before (B), at the beginning (0 min), during (20 min, 40 min), and immediately (E) after the exhaustive cycling exercise challenge.The pulmonary oxygen consumption (VO2) and carbon dioxide production (VCO2) during exercise were used to determine metabolic substrate utilization. The gaseous exchange ratio during exercise reflects the relative contributions of carbohydrates and fat to energy metabolism. The RER was calculated by dividing the VCO2 value by the VO2 value (RER =(VCO2)⁄(VO2 )). The fat oxidation rate was calculated using the following equation: Fat oxidation rate=1.695×VO2-1.701×VCO2 ). Similarly, the carbohydrate oxidation rate was calculated using the following equation: Carbohydrate oxidation rate=4.585×VCO2-3.226×VO2

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Piao Tsao, Study Chair — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsao JP, Wu PY, Kuo HT, Hong WH, Chen CC, Wang MY, Korivi M, Cheng IS. Effect of astaxanthin supplementation on cycling performance, muscle damage biomarkers and oxidative stress in young adults: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Jul 4;17(1):180. doi: 10.1186/s13102-025-01221-3. PMID 40615903